CLINICAL TRIAL: NCT00355446
Title: Bioavailabilty of Bimatoprost Ophthalmic Solution in Human Aqueous.
Brief Title: Bioavailability of Bimatoprost Ophthalmic Solution in Human Aqueous.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0106-24
Record Dates: First submitted 2006-07-20; First posted 2006-07-24 (Estimated); Last update posted 2007-10-17 (Estimated); Status verified 2007-10

CONDITIONS: Cataract
Keywords: Cataract; Human Aqueous
MeSH Terms: conditions — Cataract

INTERVENTIONS:
Drug: Bimatoprost 0.03%

SUMMARY:
The purpose of this study is to assay human aqueous for bimatoprost and the presence of any metabolites, especially prostaglandin analogs. Hypothesis:Bimatoprost is not metabolized to a prostaglandin F-2-alpha analog in human eyes

* Bimatoprost levels in human aqueous peak approximately three hours post dosing

DETAILED DESCRIPTION:
The purpose of this study is to assay human aqueous for bimatoprost and the presence of any metabolites, especially prostaglandin analogs

ELIGIBILITY:
Inclusion Criteria:

* All subjects must:

  1. Be willing and able to provide written Informed Consent.
  2. Be able and willing to follow instructions and likely to complete the entire course of the study.
  3. Be male or female of any race at least 18 years of age.
  4. Have visually significant cataract for which they have elected to undergo cataract surgery..

Exclusion Criteria:

* No subject may:

  1. Have any contraindication to use of a prostaglandin analog or prostamide derivative.

  3. Have any active ocular disease other than glaucoma or ocular hypertension that would interfere with study parameters (such as: uveitis, ocular infection, or severe dry eye). Patients with mild chronic blepharitis, age-related macular degeneration, background diabetic retinopathy may be enrolled at the discretion of the investigator.

  4. Have laser or any other intraocular surgery within the past three months. 5. Require use of ocular medications (including glaucoma medications), except intermittent use of artificial tears. Patients may not have a history of ever having used a prostaglandin analog topically.

  6. Have known allergy or sensitivity to the study medications or their components 7. Have corneal abnormalities that would interfere with the ability to obtain an adequate sample safely or have a shallow anterior which would make obtaining an aqueous sample difficult at the time of surgery in the opinion of the investigator.

  8. Be concurrently enrolled in an investigational drug or device study or participation within the last 30 days in any investigational drug or device study.

  9. Be pregnant, nursing, planning a pregnancy, or be of childbearing potential and not using a reliable form of contraception (a woman is considered of childbearing potential unless she is postmenopausal, has had a uterus and/or both ovaries removed, or has had a bilateral tubal ligation).

  10. Have a situation or condition that in the investigator's opinion may put the subject at significant risk, may confound the study results, or may interfere significantly with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2001-07; Study Completion 2004-10

PRIMARY OUTCOMES:
Bimatoprost free acid in human aqueous

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Cantor, MD, Principal Investigator — IUPUI/Clarian
Locations (4):
- United States (4):
  - University Hospital, Indianapolis, Indiana
  - Veterans Affairs Medical Center, Indianapolis, Indiana
  - Wishard Memorial Hospital, Indianapolis, Indiana
  - IU Eye at Carmel, Indianapolis, Indiana

REFERENCES:
- [Background] Cantor LB, Donnenfeld E, Katz LJ, Gee WL, Finley CD, Lakhani VK, Hoop J, Flarty K. Penetration of ofloxacin and ciprofloxacin into the aqueous humor of eyes with functioning filtering blebs: a randomized trial. Arch Ophthalmol. 2001 Sep;119(9):1254-7. doi: 10.1001/archopht.119.9.1254. PMID 11545629
- [Background] Sjoquist B, Basu S, Byding P, Bergh K, Stjernschantz J. The pharmacokinetics of a new antiglaucoma drug, latanoprost, in the rabbit. Drug Metab Dispos. 1998 Aug;26(8):745-54. PMID 9698288
- [Background] Basu S, Sjoquist B, Stjernschantz J, Resul B. Corneal permeability to and ocular metabolism of phenyl substituted prostaglandin esters in vitro. Prostaglandins Leukot Essent Fatty Acids. 1994 Apr;50(4):161-8. doi: 10.1016/0952-3278(94)90139-2. PMID 8022849